CLINICAL TRIAL: NCT04304352
Title: A Phase II Study of Metronomic Oral Chemotherapy With Cyclophosphamide Plus Capecitabine and Vinorelbine in Metastatic Breast Cancer Patients
Brief Title: Metronomic Oral Chemotherapy With Cyclophosphamide, Capecitabine and Vinorelbine in Metastatic Breast Cancer Patients
Acronym: VEX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO S582/111 RE324/2
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Vinorelbine; Capecitabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metronomic VEX (Experimental): Metronomic VEX (Oral Cyclophosphamide 50 mg daily continuous, Oral Capecitabine 500 mg, thrice daily continuous, Oral Vinorelbine 40 mg day 1,3 and 5 every week
  Interventions: Drug: Vinorelbine; Drug: Capecitabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Vinorelbine — Metronomic Vinorelbine 40 mg orally thrice a week
  Other Names: Metronomic Vinorelbine
Drug: Capecitabine — Metronomic Capecitabine 500 mg, thrice daily
  Other Names: Metronomic Capecitabine
Drug: Cyclophosphamide — Metronomic Cyclophosphamide 50 mg daily
  Other Names: Metronomic Cyclophosphamide

SUMMARY:
This is a phase II study assessing the activity and safety of metronomic chemotherapy with cyclophosphamide and capecitabine and vinorelbine in advanced breast cancer patient in four different cohort of patients:

1. Untreated (naïve) patients with endocrine responsive disease
2. Pretreated patients with endocrine responsive disease
3. Untreated (naïve) patients with triple negative disease
4. Pretreated patients with triple negative disease The primary endpoint will be the progression-free survival

DETAILED DESCRIPTION:
This is an institutional, monocentric, open-label, phase II study of oral "metronomic" Vinorelbine plus Capecitabine and Cyclophosphamide (VEX) in patients with advanced breast cancer .

Patients will receive the combination regimen as follow:

Cyclophosphamide 50 mg daily Capecitabine 500 mg, thrice daily Vinorelbine 40 mg orally thrice a week

Four independent cohorts of patients will be evaluated in the study:

1. Untreated (naïve) patients with endocrine responsive disease
2. Pretreated patients with endocrine responsive disease
3. Untreated (naïve) patients with triple negative disease
4. Pretreated patients with triple negative disease Combination will be administered until disease progression or unacceptable toxicity.

The primary endpoint will be to assess the Time to progression (TTP) of VEX combination in the four different cohorts

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or post-menopausal women (age ≥18 years) with histologically or cytologically (cell block) proven, locally advanced (inoperable) or metastatic breast carcinoma. Immunohistochemical evaluation of estrogen receptor (ER), progesterone receptor (PgR), human epidermal growth factor receptor 2 (HER2), and epidermal growth factor receptor (EGFR) according to European Institute of Oncology guidelines is mandatory.
2. Patients with HER2 overexpressed tumors, are eligible if they had received previous trastuzumab therapy for advanced disease, and/or a treatment with anti HER2 targeted therapy.
3. Patients fulfilling one of the following criteria:

   * Patients with measurable disease as per RECIST 1.1 criteria. This is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20 mm with conventional techniques or as 10 mm with spiral CT scan
   * Patients with bone lesions, lytic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST 1.1 criteria. Bone lesions must be evaluable by plain CT or MRI. Patients with lesions identified only on radionucleotide bone scan are not eligible.
4. Patients may have received any primary and/or adjuvant therapies, as any previous lines of chemotherapy and endocrine therapy for advanced disease. Patients may have received metronomic capecitabine, methotrexate and cyclophosphamide in adjuvant setting at least 12 months before study entry
5. Previous treatment with capecitabine, cyclophosphamide and vinorelbine not in metronomic schedule for advanced disease is allowed, provided that the patient has progressive disease at study entry and the patients should not be defined as "refractory" to treatments (Pathological Response or Complete Response or Stable Disease > 6 months).
6. Patients may have had previous hormonal therapy as treatment of metastatic disease provided that the patient has progressive disease at study entry. Hormonal therapy must be discontinued prior to study entry, excluding Luteinizing Hormone-Releasing Hormone (LHRH) analogue.
7. Life expectancy greater than 6 months.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status performance status <2
9. Patients must have normal organ and marrow function as defined below:

   * leukocytes ≥ 3,000/μL
   * absolute neutrophil count ≥ 1,000/μL
   * platelets ≥ 100,000/μL
   * Haemoglobin ≥ 10 g/dl
   * total bilirubin within normal institutional limits
   * Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) ≤ 2 X institutional upper limit of normal
   * creatinine within normal institutional limits OR
   * creatinine clearance ≥ 60 mL/min/1.73 m for patients with creatinine levels above institutional normal
10. Geographically accessible for follow up.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Previous metronomic chemotherapy for advanced disease with capecitabine, cyclophosphamide and vinorelbine
2. Patients defined as "refractory" to capecitabine, cyclophosphamide and vinorelbine (Progression Disease or Stable Disease < 6 months).
3. Presence of symptomatic cerebral or leptomeningeal involvement.
4. Previous or concomitant other malignancy except basal or squamous cell carcinoma of the skin or adequately treated in situ carcinoma of the cervix.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Malabsorption syndrome or disease affecting significantly gastrointestinal function or major resection of the stomach or proximal small bowel that could affect absorption of oral vinorelbine
7. Concurrent treatment with any other anti-cancer therapy except LHRH analogue.
8. Patients with pre-existing motor or sensory peripheral neuropathy grade 2 according to NCI criteria

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2011-07-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | 28 days
  the time between the first study dose administration and the date of progression of the disease or cancer-related death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Marco Colleoni, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No